CLINICAL TRIAL: NCT03295188
Title: A Randomized Double-Blind Placebo-Controlled Study to Evaluate the Effects of Scallop-derived Plasmalogen on Obese Subjects
Brief Title: Effects of Plasmalogen on Obese Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Japanese Plasmalogen Society (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pls2017-01
Record Dates: First submitted 2017-09-24; First posted 2017-09-27 (Actual); Last update posted 2019-02-19 (Actual); Status verified 2019-02

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Plasmalogens

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Two 0.5 mg plasmalogen capsules per day
  Interventions: Dietary Supplement: Plasmalogen
- Placebo Group (Placebo Comparator): Two placebo capsules containing no plasmalogen per day
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Plasmalogen — Treatment group takes two 0.5 mg plasmalogen capsules per day for 12 weeks.
  Arms: Intervention Group
Dietary Supplement: Placebo — Placebo Group takes two placebo capsules per day for 12 weeks.
  Arms: Placebo Group

SUMMARY:
This is a 12-week, randomized, double-blind, placebo-controlled study to evaluate the effects of scallop-derived plasmalogen on brain fatigue, body weight and changes in blood plasmalogen in obese subjects aged 20-75 years old.

ELIGIBILITY:
Inclusion Criteria:

* Willingness to provide informed consent to participate in the study
* BMI ≥ 25 ㎏/㎡
* HbA1C ≺ 8% without antidiabetic medication in the previous 3 months
* Stable medication for 3 months prior to the enrollment, and expectedly throughout the course of study

Exclusion Criteria:

* Scallop allergy
* Symptomatic obesity, i.e., endocrinal, hypothalamic or drug-induced obesity
* Hypertension under medication with 4 or more drugs
* Hepatic disorder with AST ≥ 5 times upper limit of the normal range
* Mental disorder including schizophrenia and neurosis
* Alcohol dependence
* History of malignancy for which treatment completed in the past 5 years
* Inflammatory disease
* Use of plasmalogen supplement in the past 3 months
* Ineligible condition as determined by study physician

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2017-12-08 (Actual); Primary Completion 2018-08-22 (Actual); Study Completion 2018-08-22 (Actual)

PRIMARY OUTCOMES:
Change in Profile of Mood States 2nd Edition (POMS 2) | 12 weeks
  Psychological rating scale to assess transient feelings and mood

SECONDARY OUTCOMES:
Change in body weight | 12 weeks
Change in waist diameter | 12 weeks
Change in blood levels of plasmalogen | 12 weeks
Change in Athens Insomnia Scale (AIS) | 12 weeks
  Self-assessment psychometric tool to quantify sleep difficulty
Changes in adiponectin, leptin, IRI, GA, and high sensitive quantitation of C-reactive protein | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Takehiko Fujino, Study Chair — BOOCS Clinic Fukuoka
Locations (1):
- BOOCS Clinic Fukuoka, Fukuoka, Japan